CLINICAL TRIAL: NCT06527014
Title: Comparison of the Effectiveness of Pulsed Radiofrequency (pRF) to the Suprascapular Nerve Versus Conventional Physical Therapy Program in Chronic Shoulder Pain
Brief Title: Pulsed Radiofrequency to the Suprascapular Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hüma Bölük Şenlikci, Associate Professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent1
Record Dates: First submitted 2024-07-21; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic; Shoulder Pain
Keywords: Pain; Injections; Nerve Block; Shoulder pain; Function
MeSH Terms: conditions — Chronic Pain; Shoulder Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulse Radiofrequency-Group 1 (Active Comparator): Procedures were performed with patient seated leaving their affected shoulder exposed. First, the spina scapula was identified and scapular notch and transverse scapular ligament identified. The needle was inserted out plane. A standard radiofrequency device (NeuroTherm NT1100, Neurotherm Inc.,USA) was used with 22-gauge 10-cm, 5 mm RF cannulas (Abbott Medical , USA) for SN blocks.The cannula was placed through the transverse scapular ligament area and sensory fibre stimulation was started between 0.3 and 1 V. The patient was asked for feedback on symptoms such as numbness, paresthesia and/or pain. If the patient did not report any sensory symptoms within the specified sensory stimulation range, the cannula was repositioned. Motor stimulation was applied up to 2 V and it was checked whether there was any muscle contraction or not. If any contraction was figured out as a result of motor stimulation.Eventually, the SN was ablated at 42°C for 4 minutes in pRF mode.
  Interventions: Procedure: Pulse Radiofrequency to the suprascapular nerve
- Conventional Physical Therapy-Group 2 (No Intervention): Patients in the Group 2 received physical therapy modalities including hot packs, transcutaneous electrical nerve stimulation (TENS) and deep heater ultrasound to the shoulder. The hot packs were preserved at 71°C, then application of hot packs were done at a temperature of 40-43°C with TENS (4 cannulated electrodes) adjusted at 60-100 Hz for 20 minutes. Therapeutic deep heater ultrasound was applied to warm up subcutaneous tissues for 10 minutes at 1.5 watts/cm2. Until follow-up process was over, no medications other than paracetamol were allowed.

INTERVENTIONS:
Procedure: Pulse Radiofrequency to the suprascapular nerve — Pulse radiofrequency ablation to the Suprascapular nerve
  Arms: Pulse Radiofrequency-Group 1

SUMMARY:
Regardless of the etiology, chronic shoulder pain is a distressing condition that affects daily life and is among the first common reasons for musculoskeletal system problems when admitting to clinics. Pulsed radiofrequency (pRF) treatment to the suprascapular nerve (SSN) is a promising interventional procedure, that is thought to be effective in case of chronic shoulder pain. However, conventional physical therapy program is preferred more often and found more applicable. The aim of current study is to compare the effectiveness of two treatment procedures.

DETAILED DESCRIPTION:
This study carried out in 27 chronic shoulder pain patients aged between 18-75 years in Ankara Bilkent City Hospital, Physical Medicine and Rehabilitation Hospital. Total of 25 patients, who had > 3 months shoulder pain and pain more than > 4 according to the numerical rating scale (NRS), completed the study. Twenty-seven patients randomized into two groups, 21 patients underwent pRF of Suprascapular nerve (SSN) in Group 1; 16 patients received 10 sessions conventional physical therapy (CPT) program. One patient did not come to follow-ups after SSN pRF procedure, other patient did not complete the 10 session CPT program.

Approval for the study was granted by the 2nd Ethics Committee of Ankara Bilkent City Hospital (Protocol number: E2-23-3799). The study was conducted in line with the Helsinki Declaration. All patients signed informed consent prior to participation.

Inclusion criteria were 1) shoulder pain lasts more than 3 months 2) Shoulder pain more than 4 according to NRS 3) no passive range of motion limitation 4) unilateral chronic shoulder pain 5) INR> 1.2 in blood samples.

Exclusion criteria were 1) Adhesive capsulitis that cause passive range of motion in shoulder joint 2) History of intra-articular joint injection or physical therapy at the last 6 months 3) History of fracture, trauma or surgery 4) Accompanying rheumatologic disease or other inflammatory arthritis involved shoulder joint 5) Local infection, sepsis, malignancy or pregnancy 6) Uncontrolled diabetes or other co-morbidities that worsens general condition 7) History of allergy to the materials used in treatment 8) Mental disorders that lead incooperation.

After the informed consent patients divided into 2 groups with closed envelope method by the staff who is not participated in the study. Group 1 underwent SSN pRF and Group 2 received 10 sessions of CPT program including hotpack, therapeatic ultrasound as a deep heater and transcutaneous electrical nerve stimulation (TENS). All patients were thought shoulder exercises such as pendulum exercises and isometric exercises around shoulder muscles to be performed individually until the 1st month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain lasts more than 3 months
* Shoulder pain more than 4 according to NRS
* No passive range of motion limitation
* Unilateral chronic shoulder pain
* INR> 1.2 in blood samples.

Exclusion Criteria

* Adhesive capsulitis that cause passive range of motion in shoulder joint
* History of intra-articular joint injection or physical therapy at the last 6 months
* History of fracture, trauma or surgery
* Accompanying rheumatologic disease or other inflammatory arthritis involved shoulder joint
* Local infection, sepsis, malignancy or pregnancy
* Uncontrolled diabetes or other co-morbidities that worsens general condition
* History of allergy to the materials used in treatment
* Mental disorders that lead incooperation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Numarical Rating Scale | partcipants were evaluated at baseline and 1st month follow-up
  Numerical rating scale (NRS): It is a rating scale for self reported pain. 0 , means there is no pain and 10, represents the most pain experienced in life time.
QuickDASH | partcipants were evaluated at baseline and 1st month follow-up
  It is self-reported questionnaire related to pain and disfunction. Abilities and symptoms are asked about last week. All questions are rated 0-5. Higher scores are related more disability for upper extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Adıgüzel, Prof, Study Chair — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bİlkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data is going to be shared after review process

REFERENCES:
- [Result] Akbari N, Ozen S, Senlikci HB, Haberal M, Cetin N. Ultrasound-guided versus blind subacromial corticosteroid and local anesthetic injection in the treatment of subacromial impingement syndrome: A randomized study of efficacy. Jt Dis Relat Surg. 2020;31(1):115-22. doi: 10.5606/ehc.2020.71056. PMID 32160504
- [Result] Crookes T, Wall C, Byrnes J, Johnson T, Gill D. Chronic shoulder pain. Aust J Gen Pract. 2023 Nov;52(11):753-758. doi: 10.31128/AJGP-04-23-6790. PMID 37935145
- [Result] Esparza-Minana JM, Mazzinari G. Adaptation of an Ultrasound-Guided Technique for Pulsed Radiofrequency on Axillary and Suprascapular Nerves in the Treatment of Shoulder Pain. Pain Med. 2019 Aug 1;20(8):1547-1550. doi: 10.1093/pm/pny311. PMID 30690499
- [Result] Bergamaschi ECQA, Sakata RK, Giraldes ALA, Ferraro LHC. Comparative Randomized Study Between Pulsed Radiofrequency and Suprascapular Nerve Block for the Treatment of Chronic Shoulder Pain. Clin J Pain. 2024 Mar 1;40(3):182-186. doi: 10.1097/AJP.0000000000001184. PMID 38050367